CLINICAL TRIAL: NCT05127655
Title: Assessment of Oral Health Related Quality of Life After Full Mouth Rehabilitation Under General Anesthesia in a Group of Egyptian Children Below 5 Years Old (A Before and After Study)
Brief Title: Assessment of Oral Health Related Quality of Life After Full Mouth Rehabilitation Under GA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eyman Sheikh Eldin Mokhtar, Doctor Eyman sheikh eldin mokhtar pedodontist principle investigator, Cairo University
Other Study IDs: OHRQOL in 5 years children
Record Dates: First submitted 2018-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Quality of Life
Keywords: Rehabilitation; full mouth rehabilitation; Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: full mouth rehabilitation — full mouth rehabilitation under general anesthesia

SUMMARY:
To assess Oral health related quality of life (OHRQOL) after full mouth rehabilitation under GA in a group of Egyptian children below 5 years

ELIGIBILITY:
Inclusion Criteria:

* Age range 2 to 5 years .
* Children with untreated early childhood caries .
* Children who will undergo dental treatment under general anesthesia.

Exclusion Criteria:

* Participation in any other concurrent clinical trials.
* The presence of serious medical conditions or a transmissible disease such as malignant disease, hepatitis, AIDS etc.
* Children with special healthcare needs.
* Children whose parents had no home or mobile phone to enable postoperative contact.
* Parent that will not sign the consent.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Caregivers paired with their children attending Pediatric Dentistry and Dental Public Health department, faculty of dentistry, Cairo University Egypt
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Oral health related quality of life (OHRQOL) | change from baseline oral health related quality of life at 6 months
  Oral health related quality of life (OHRQOL) will be measured by validated questionnaire which is : Early Childhood Oral Health Impact Scale (ECOHIS) .
  the unit of measurement is likert scale.

SECONDARY OUTCOMES:
Body mass index | change of baseline body mass at 6 months
  Children's weights will be measured in kilograms and heights in meters .Body max index (BMI) will be calculated using this formula: BMI = weight (kg) / height (m)² to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Korany, PHD, Study Director — Cairo University